CLINICAL TRIAL: NCT03983772
Title: A Pilot Study to Evaluate the Gastrointestinal Response to Increasing Doses of a Resistant Starch Blend in Healthy Subjects
Brief Title: Resistant Starch Blend Gastrointestinal Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Collaborators: Personalized Lifestyle Medicine Center (Unknown); National University of Natural Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RSBGI-PLMC
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Quality of Life; Health, Subjective
Keywords: Prebiotics; Resistant starch; Gut microbiota; Microbial diversity; Dietary fiber; Short-chain fatty acid; Gastrointestinal symptom; Dose-ramping design; Resistant starch blend; Fecal consistency; Fecal frequency; PROMIS; Microbiome analysis; Virtual; Remote access

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind (subject)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RS10-10-10 (Experimental): First 2 weeks is for baseline variability measurement (no product). Second 2 weeks is 10 g resistant starch (RS) blend. Third 2 weeks is 10 g RS blend. Fourth 2 weeks is 10 g RS blend.
  Interventions: Dietary Supplement: RS blend
- RS10-20-20 (Experimental): First 2 weeks are for baseline variability measurement (no product). Second 2 weeks is 10 g resistant starch (RS) blend. Third 2 weeks is 20 g RS blend. Fourth 2 weeks is 20 g RS blend.
  Interventions: Dietary Supplement: RS blend
- RS10-20-30 (Experimental): First 2 weeks are for baseline variability measurement (no product). Second 2 weeks is 10 g resistant starch (RS) blend. Third 2 weeks is 20 g RS blend. Fourth 2 weeks is 30 g RS blend.
  Interventions: Dietary Supplement: RS blend
- Placebo10-10-10 (Placebo Comparator): First 2 weeks are for baseline variability measurement (no product). Second 2 weeks is 10 g placebo. Third 2 weeks is 10 g placebo. Fourth 2 weeks is 10 g placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: RS blend — The intervention is a proprietary resistant starch blend.
  Arms: RS10-10-10; RS10-20-20; RS10-20-30
Other: Placebo — The placebo is starch.
  Arms: Placebo10-10-10

SUMMARY:
This study aims to test the hypothesis that a unique blend of resistant starches and fiber will promote gastrointestinal health, as measured by an increase in short-chain fatty acids and improvement in quality of life measures in conjunction with microbial community changes. This study specifically evaluates the impact on short-chain fatty acids and gut microbiota and the impact on quality of life from a resistant starch blend in healthy adult humans with occasional gastrointestinal distress.

DETAILED DESCRIPTION:
Low microbial diversity in the intestine correlates with chronic diseases such as Inflammatory Bowel diseases, colorectal cancer, obesity, Type 1 and Type 2 diabetes and more. The incidence of chronic diseases is greater in the industrialized society consuming a diet low in microbiota-accessible-carbohydrates. Thus, research is growing to seek prebiotics, which are substrates that host microbes selectively use, providing a health benefit.

Better-tolerated prebiotics may be desirable, particularly for those avoiding FODMAPs (fermentable oligosaccharides, disaccharides, monosaccharides and polyols) due to gastrointestinal distress. Additionally, the intestinal microbiome may benefit from a diversity of prebiotics that may affect different types of bacteria to contribute to overall microbial diversity as well as provide stronger effects on positive outcomes. Resistant starch type 2, also called RS2, so named due to its ability to resist digestion in the upper gastrointestinal tract, is a candidate prebiotic, growing in popularity for increasing beneficial intestinal bacteria and improving gastrointestinal symptoms and reducing glycemic responses.

This study aims to test the hypothesis that a unique blend of resistant starches and fiber will promote gastrointestinal health, as measured by an increase in short-chain fatty acids and improvement in quality of life measures in conjunction with microbial community changes. This study specifically evaluates the impact on short-chain fatty acids and gut microbiota and the impact on quality of life from a resistant starch blend in healthy adult humans with occasional gastrointestinal distress.

ELIGIBILITY:
* Willingness to maintain current lifestyle (diet and exercise) practices (other than avoiding or limiting alcohol)
* Willing to avoid alcohol during the study OR limit alcohol consumption to 1-2 glasses of light beer or wine for the 1-2 days after the stool collection for visits 2, 3 and 4 (Participants who choose to consume alcohol will be given List of Foods A and Participant Checklist A while others will be given the B versions)
* Willingness to give informed consent to participate in the study.
* Presence of minor symptoms of bloating or constipation or irregular bowel movements
* Willingness and ability to collect per the two stool test kit procedures 10 stool samples at home and ship per instructions
* Willing to have blood drawn 3 times (not applicable to those impacted by circumstances associated with COVID-19 pandemic)
* Ability to speak, read and understand English
* Ability to participate via telemedicine (phone or video calls for study visits and submit documents electronically and receive products and return unused products)

Exclusion criteria 4.1.1 Prohibited Medications, Supplements or Herbal Products Exclusionary

* Currently taking a probiotic, resistant starch, prebiotic or fiber supplement (or they were taken within the last 14 days)
* Currently taking antibiotic, antiparasitic, or antifungal medications orally or intravenously (or they were taken within the last 28 days)
* Initiation of/or changes to supplements or medications within 28 days prior to screening
* Currently taking any supplements or medications impacting gastrointestinal motility (e.g., SSRI's, PPI's, opioids) (one exception is use of PPI's if the PPI use is stable, i.e., dosage and frequency is consistent, has not changed in the last month, and will not change during the course of the study. Such individuals may be included in the study at the discretion of the investigator)
* The use of any supplements or medications which influences digestion and absorption of nutrients

4.1.2 Medical History and Concurrent Diseases Exclusions

* No serious, unstable illnesses including cardiovascular, hepatic, renal, gastrointestinal, respiratory, endocrine, neurologic, immunologic, or hematologic disease.
* Known infection with Human Immunodeficiency Virus (HIV), Tuberculosis or Hepatitis B or C.
* Known intolerance or allergy to ingredients in test study product
* Active and severe gastrointestinal symptoms and/or infections
* The presence of any disease which influences digestion and absorption of nutrients
* History of any bariatric surgery procedure within the last 5 years
* History of gastrointestinal surgery within the last 5 years
* Currently have a colostomy or ileostomy bag in place
* Genito-urinary bacterial infections within the last 28 days
* Any cardiovascular disease including myocardial infarction, angina, cardiovascular surgery, congestive heart failure, cardiac arrhythmias or conduction abnormalities, cerebrovascular accident, transient ischemic attack (TIA), or peripheral vascular disease, deep vein thrombosis or pulmonary embolus.
* Any personal history of pre-Diabetes, Diabetes Mellitus Type 1 or 2 or hypoglycemia.
* Personal history of seizure disorder other than a single childhood febrile seizure that fully resolved.
* Any personal history of bipolar disorders, schizophrenia or psychotic behaviors.
* Any serious mental illness including depression, manic episodes, post-traumatic disorder, obsessive-compulsive disorder, personality disorders, history of attempted suicide or violence within 12 months prior to Screening and for the duration of the study.
* A major medical or surgical event requiring hospitalization (for any reason other than a scheduled medical procedure) within the preceding 3 months
* Malignancy within the last 5 years (with the exception of basal cell carcinoma, squamous cell carcinoma, and/or carcinoma in situ of the cervix)
* Women who are lactating, pregnant or planning pregnancy within the next three months 4.1.3 Substance Use Exclusions
* Smoking or use of nicotine containing products 30 days prior to Screening and for the duration of the study.
* History of alcohol abuse or a diagnosis of alcoholism within 12 months prior to Screening and for the duration of the study.
* Consumption of alcohol (or more than 4 glasses within the last 2 weeks if considered for the light alcohol use category, and no more than 2 glasses at once) for 14 days prior to Screening.
* Use of drugs of abuse and recreational drugs/substances (such as but not limited to opioids, cocaine, phencyclidine [PCP], and methamphetamine, including marijuana or cannabinoids) within 12 months prior to Screening and for the duration of the study.

4.1.4 Other Exclusionary Criteria

* Inability to comply with study and/or follow-up visits.
* Any other concurrent condition which, in the opinion of the Investigator, would preclude participation in this study or interfere with compliance.
* Initiation of or changes to an exercise regimen within 28 days prior to screening
* Initiation of or changes to a food plan within 28 days prior to screening
* Current involvement or within 28 days prior to screening of a significant diet or weight loss program, such as NutriSystem, Jenny Craig, Atkin's or other low-carb diet programs, or very low calorie liquid diet programs (such as Optifast, Medifast, and/or HMR) or any diet that has led to a weight loss of 5% of body weight over a period of 10 weeks.
* Difficulty or aversion to taking powdered supplement
* Currently participating in another interventional research study or participated in another interventional study within the previous 28 days

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Concentration of short-chain fatty acids from baseline to each product intervention | Baseline (2 week period) compared to each product completion period of 2 weeks
  Concentration of total short-chain fatty acids, including valerate, isovalerate and isobutyrate, and individually-reported n-butyrate concentration as well as propionate and acetate % will be reported by Genova Diagnostics Report

SECONDARY OUTCOMES:
Change in fecal frequency (hours between stools) from baseline at each intervention | Baseline (2 week period) to end of product completion (2 week intervention for each dose and time combination)
  Fecal frequency (time in hours between stools) will be evaluated for each time period and compared between baseline (2 week period) and product intervention period (each 2 week period)
Change in Response pattern score for Frequency and Severity of Gastrointestinal Symptoms (PROMIS Scale v1.0 - GI Diarrhea 6a) | Baseline (2 week period) to end of product completion (2 week intervention for each dose and time combination)
  Response pattern score on PROMIS Scale v1.0 - GI Diarrhea will be compared between baseline and each intervention period
Change in Response pattern score for Frequency and Severity of Gastrointestinal Symptoms (PROMIS Scale v1.0 - GI Constipation) | Baseline (2 week period) to end of product completion (2 week intervention for each dose and time combination)
  Response pattern score on PROMIS Scale v1.0 - GI Constipation will be compared between baseline and each intervention period
Change in Response pattern score for Frequency and Severity of Gastrointestinal Symptoms (PROMIS Scale v1.0 - GI Gas and Bloating 13a 09-02-2016) | Baseline (2 week period) to end of product completion (2 week intervention for each dose and time combination)
  Response pattern score on PROMIS Scale v1.0 - GI Gas and Bloating 13a 09-02-2016 will be compared between baseline and each intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Patno, PhD, Principal Investigator — Metagenics, Inc.; Joseph Lamb, MD, Principal Investigator — PLMC
Locations (1):
- Personalized Lifestyle Medicine Center, Gig Harbor, Washington, United States

IPD SHARING:
Plan to Share IPD: No